CLINICAL TRIAL: NCT05717426
Title: The Effects of Open Versus Closed Kinetic Chain Exercises on Ankle Joint Function in Athletes With Chronic Ankle Instability
Brief Title: The Effects of Open Versus Closed Kinetic Chain Exercises on Ankle Joint Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ahmadsajjad0446
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open chain exercises group (Active Comparator): Group A(Open chain exercises group) received open kinetic exercises 3 times a week for 3-4 weeks.
  Interventions: Other: Open chain exercises
- Closed kinetic chain exercises group (Active Comparator): Group B(Closed kinetic chain exercises group) received close kinetic exercises 3 times a week for 3-4 weeks.
  Interventions: Other: Closed kinetic chain exercises

INTERVENTIONS:
Other: Open chain exercises — An open chain exercise is one that allows the furthest part of the chain to move freely. For example, picking up a glass of water is an open-chain exercise. The hand affects the elbow and the shoulder as it is not fixed in place. However, it does not effect the rest of your body.
  Arms: Open chain exercises group
Other: Closed kinetic chain exercises — Closed Kinetic Chain (CKC) exercises or closed chain exercises are exercises or movements where the distal aspect of the extremity is fixed to an object that is stationary.
  Arms: Closed kinetic chain exercises group

SUMMARY:
The goal of this Randomized clinical trial is to find the effects of open versus closed kinetic chain exercises on ankle joint function in athletes with chronic ankle instability. The main question it aims to answer is:

• To compare the effects of open versus closed kinetic chain exercises on pain, instability and balance in athletes with chronic ankle instability.

Participants were given consent form and after subjects read and signed the informed consent and completed the self-reported questionnaires designed to identify subjects with CHRONIC ANKLE INSTABILITY, subjects completed baseline measurements that included Foot and Ankle Ability Measure (FAAM)-Sport Subscale, Reach distance, and SEBT. Participant were divided into two groups (Group A and Group B) through lottery method. Group A received open kinetic exercises 3times a week for 3-4 weeks. Group B received close kinetic exercises 3 times a week for 3-4 weeks.

DETAILED DESCRIPTION:
Chronic instability is a common condition in sports and there are many treatment methods and rehabilitation protocols available which are used according to extent of injury. The purpose of this study is to find out the effects of close kinetic chain exercises and open kinetic chain exercises and to find out which technique is more efficient for treating ankle instability, pain, and imbalance in athletes with chronic ankle instability. This study will help physical therapists and medical team to enhance the rehabilitation process.

The study was randomized clinical trial conducted at Pakistan Sports board Lahore in which convenient random sampling technique was used. This study included total 26 participants and for this purpose Open Epi tool would be used as a sample size calculation. Participants falling in this category were recruited into the study after inclusion and exclusion criteria. The Cumberland ankle instability tool was used as a tool for pre and post assessment of athletes. In this study we divided population into two groups. Group A received open chain kinetic exercises and Group B was treated with Closed chain kinetic exercises. Data was analyzed through SPSS 25 version.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-30years
* Tennis, Football, Cricketers, volley ball and Hockey players
* Athletes with balance problems
* Chronic ankle injuries

Exclusion Criteria:

* Acute injuries
* Non-athletes (minimum once a week sports participation)
* Athletes with pain related to calf muscles and achillies tendon

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4 weeks
  The Numeric Pain Rating Scale (NPRS) is commonly used to assess pain. Change in the NPRS across time can be interpreted with responsiveness indices.
Star excursion balance test. | 4 weeks
  The SEBTs are functional tests that incorporate a single-leg stance on one leg with maximum reach of the opposite leg. The SEBTs are performed with the subject standing at the center of a grid placed on the floor, with 8 lines extending at 45° increments from the center of the grid. The 8 lines positioned on the grid are labeled according to the direction of excursion relative to the stance leg: anterolateral (AL), anterior (A), anteromedial (AM), medial (M), posteromedial (PM), posterior (P), posterolateral (PL), and lateral (L). The grid was constructed in an athletic training facility using a protractor and 3-in (7.62-cm)-wide adhesive tape and was enclosed in a 182.9-cm by 182.9-cm square on the hard tile floor.
Reach distance. (functional reach test) | 4 weeks
  Functional Reach (standing instructions): The patient is instructed to next to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the starting position at the 3rd metacarpal head on the yardstick. Instruct the patient to "Reach as far as you can forward without taking a step." The location of the 3rd metacarpal is recorded. Scores are determined by assessing the difference between the start and end position is the reach distance, usually measured in inches. Three trials are done and the average of the last two is noted.
Cumberland Ankle Instability Tool (CHRONIC ANKLE INSTABILITYT) and Ankle Instability Instrument (AII) | 4 weeks
  The Cumberland Ankle Instability Tool (CHRONIC ANKLE INSTABILITYT) is a PROM that can detect functional ankle instability and provide a measure of the severity of the instability . It does so through nine questions evaluating ankle pain, subjective instability during activities such as running or hopping and the ability of the ankle to cope with episodes of giving way . The answers for the nine questions are added up to a total score, which goes from 0 (indicating an extreme functional instability of the ankle) to 30 points (indicating a stable ankle)
Foot and Ankle Ability Measure (FAAM)-Sport Subscale | 4 weeks
  The Foot and Ankle Ability Measure (FAAM) is a patient-reported questionnaire for patients with muscu loskeletal foot and ankle disorders consisting of two sub scales, ADL and Sports, with a total of 32 questions. The FAAM is an evaluative self-reported instrument to comprehensively assess physical function of individu als with musculoskeletal disorders of the foot and ankle. It consists of an ADL (FAAM-ADL) and Sports (FAAM-Sport) subscale, containing 21 and 9 items, respectively. Standardized answer options are given in five-point Likert boxes, ranging from 0 (no difficulty at all) to 4 (unable to do). The sixth option is 'not applicable, which will not be taken into account when counting the percentage scores. According to Martin et al. we only calculated a total subscale if ≤2 items were missing (or inapplicable) in the FAAM-ADL and if ≤1 item was missing (or inapplicable) in the FAAM-Sport domain. A higher score represents a higher level of function in each subscale

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ahmed sajjad, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board Lahore, Lahore, Punjab Province, Pakistan